CLINICAL TRIAL: NCT00519038
Title: Experimental Prospective Study on the Effectiveness and Efficiency of the Implementation of Clinical Pathways
Acronym: EPSEEIC2004
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agenzia Regionale Sanitaria delle Marche (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EPSEEIC2004-EXART12MARCHE
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Congestive Heart Failure
Keywords: Critical Pathways; Congestive Heart Failure; Randomized Controlled Trial; Effectiveness
MeSH Terms: conditions — Heart Failure | interventions — Critical Pathways

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients treated according to clinical pathways
  Interventions: Other: Clinical Pathways
- 2 (Other): Patients treated according to usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Clinical Pathways — Clinical pathways are a methodology for the mutual decision making and organization of care for a well-defined group of patients during a well-defined period with the aim to enhance the quality of care by improving patient outcomes, promoting patient safety, increasing patient satisfaction, and optimizing the use of resources. They are also developed by multi-professional teams
  Arms: 1
Other: Usual Care — Usual care is the current practice actually performed in the hospital
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the use of clinical pathways improves the quality of the hospital care of decompensated heart failure patients.

DETAILED DESCRIPTION:
In Europe approximately 5% of all acute medical admissions relate to heart failure and in the United States heart failure is responsible for almost 1 million hospitalizations annually. Almost three quarters of these admissions are unplanned and worsening heart failure is responsible for half of these admissions.

The Acute Decompensated Heart Failure National Registry (ADHERE) showed that the hospital treatment of heart failure frequently does not follow published guidelines or conform to the Joint Commission on Accreditation of Healthcare Organizations (JCAHO) core performance measures, potentially contributing to the high morbidity, mortality and economic cost of this disorder. ADHERE findings also suggested that the wide variations in conformity may reflect differences in training, guideline familiarity, and implementation of tools and systems to ensure that recommended care is provided and documented. Consequently the development of educational and quality improvement programs has the potential to considerably reduce the current variability in care, enhance guideline adherence, and improve outcomes for patients.

Clinical pathways has become a popular tool to achieve such goals. Clinical pathways are a methodology for the mutual decision making and organization of care for a well-defined group of patients during a well-defined period with the aim to enhance the quality of care by improving patient outcomes, promoting patient safety, increasing patient satisfaction, and optimizing the use of resources. They are also developed by multi-professional teams. Despite enthusiasm and diffusion, the widespread acceptance of clinical pathways remain questionable because very little prospective controlled data demonstrated their effectiveness.

The Experimental Prospective Study on the Effectiveness and Efficiency of the Implementation of Clinical Pathways was designed in order to conduct a rigorous evaluation of a clinical pathway in hospital treatment of decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* principal diagnosis of heart failure (all ICD-9 codes included in 428.xx code)

Exclusion Criteria:

* current acute myocardial infarction (AMI)
* current unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2003-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | during the stay

SECONDARY OUTCOMES:
Appropriateness of the stay; Rate of unscheduled readmissions; Length of the stay; Cost of the admission; Patients' satisfaction score; Use of diagnostic procedures; Use of medical treatments. | during the stay or at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Gardini, MD, Study Chair — Agenzia Regionale Sanitaria delle Marche

REFERENCES:
- [Derived] Panella M, Marchisio S, Demarchi ML, Manzoli L, Di Stanislao F. Reduced in-hospital mortality for heart failure with clinical pathways: the results of a cluster randomised controlled trial. Qual Saf Health Care. 2009 Oct;18(5):369-73. doi: 10.1136/qshc.2008.026559. PMID 19812099
- [Derived] Panella M, Marchisio S, Gardini A, Di Stanislao F. A cluster randomized controlled trial of a clinical pathway for hospital treatment of heart failure: study design and population. BMC Health Serv Res. 2007 Nov 7;7:179. doi: 10.1186/1472-6963-7-179. PMID 17986361